CLINICAL TRIAL: NCT06394557
Title: Evaluation of In-office Bleaching-induced Sensitivity With 2 or 7 Days Interval Between Sessions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: In-office bleach 48h interval
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-04

CONDITIONS: Tooth Sensitivity
Keywords: dental bleaching; dentine sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bleaching 7 days interval (Active Comparator): Participants will undergo 2 sessions of in-office dental bleaching, using a 35% Hydrogen Peroxide bleaching gel, with 7 days of interval between sessions. Bleaching gel will be used in 3 15-minutes applications as indicated by the manufacturer. A 2% Potassium Nitrate and Sodium Fluoride desensitizing gel will be applied 15 minutes before the dental bleaching procedure, in both sessions.
  Interventions: Procedure: In-office Dental Bleaching Conventional
- Bleaching 2 days interval (Experimental): Participants will undergo 2 sessions of in-office dental bleaching, using a 35% Hydrogen Peroxide bleaching gel, with 2 days of interval between sessions. Bleaching gel will be used in 3 15-minutes applications as indicated by the manufacturer. A 2% Potassium Nitrate and Sodium Fluoride desensitizing gel will be applied 15 minutes before the dental bleaching procedure, in both sessions.
  Interventions: Procedure: In-office Dental Bleaching Alternative

INTERVENTIONS:
Procedure: In-office Dental Bleaching Conventional — Participants will undergo 2 sessions of in-office dental bleaching, using a 35% Hydrogen Peroxide bleaching gel, with 7 days of interval between sessions. Bleaching gel will be used in 3 15-minutes applications as indicated by the manufacturer. A 2% Potassium Nitrate and Sodium Fluoride desensitizing gel will be applied 15 minutes before the dental bleaching procedure, in both sessions.
  Arms: Bleaching 7 days interval
Procedure: In-office Dental Bleaching Alternative — Participants will undergo 2 sessions of in-office dental bleaching, using a 35% Hydrogen Peroxide bleaching gel, with 2 days of interval between sessions. Bleaching gel will be used in 3 15-minutes applications as indicated by the manufacturer. A 2% Potassium Nitrate and Sodium Fluoride desensitizing gel will be applied 15 minutes before the dental bleaching procedure, in both sessions.
  Arms: Bleaching 2 days interval

SUMMARY:
Clinical randomized single-blind trial, used to measure the level of tooth sensitivity (TS) after in-office dental bleaching sessions, on volunteers using a modified visual analog scale (VAS). The investigators selected for this study, 47 participants with color 2M2 or darker (Using 0M1 - 5M3 Vita bleaching shade guide). The investigators performed two bleaching sessions with an acidic 35% hydrogen peroxide gel with either a 1-week or 2-day interval. The investigators recorded the TS up to 48 h with a VAS scale and the color at baseline and 30 days after bleaching with a value-oriented shade guide and a spectrophotometer. The risk and intensity of TS and the color change were compared between the two groups.

DETAILED DESCRIPTION:
Two weeks before the bleaching procedures, selected volunteers from the city of Nova Friburgo, (Rio de Janeiro, Brazil) received a dental screening and a dental prophylaxis with pumice and water in a rubber cup and signed an informed consent form.

This was a randomized, single-blind (evaluators), parallel and equivalence trial with an equal allocation rate between groups.

A total of 61 participants were examined in a dental chair to check if they met the inclusion and exclusion criteria. A total of 47 participants were included in this study. The participants were randomly divided in the 2-day and 7-day groups.

During the in-office sessions, participants had the gingival tissue isolated of the teeth using a light-cured resin dam (Top Dam, FGM, Joinville, SC, Brazil). After that, a 2% Potassium nitrate and Sodium fluoride desensitizer gel (Desensitize 2%, FGM) was applied for 15 minutes before dental bleaching. This gel was removed and the 35% hydrogen peroxide gel (Whiteness HP, FGM, Joinville, Brazil) was applied in three 15-min applications according to the manufacturer's directions in all upper and lower incisors, canines and premolars. After 2 days (2-day group) and 7 days (7-day group), this procedure was repeated using the same protocol.

Color evaluation was performed before and 30 days after the end of the bleaching treatment using a subjective (value oriented shade guide Vita Lumin, Vita Zahnfabrik, Bad Sackingen, Germany) and an objective method (Easyshade spectrophotometer, Vident, Brea, CA, USA). Color evaluation was done in a room under artificial lightning conditions without interference from outside light.

For the subjective examination, the shadeguide's 16 tabs were arranged from highest (B1) to lowest (C4) value. Changes in the scale were treated as representing a continuous and approximately linear ranking. Color was measured in the middle third of the facial surface of the right upper canine at baseline and 30 days after bleaching to calculate the variations in color towards the lighter end of the scale (Delta Shade Guide Units - DSGU).

One calibrated operator measured the colour in all participants using the Vita Easyshade spectrophotomer (Easyshade, Vident, Brea, CA, USA) before and 30 days after the bleaching therapy. The L*, a* and b* parameters were recorded. L* represents the value from 0 (black) to 100 (white) and a* and b* represent the shade, where a* is the measurement along the red-green axis and b* is the measurement along the yellow-blue axis. Color change was calculated between the two assessment periods (DE) using the formula: DE = [(DL*)2 + (Da*)2 + (Db*)2]1/2.

The patients recorded their perception of TS during the first and second bleaching sessions using the visual analogue scale VAS. This scale employs a 10-cm horizontal line with words ''no pain'' at one end and ''worst pain'' at the opposite end. Participants recorded whether they experienced TS during the treatment up to 1 h after the bleaching, from 1 h to 24 h and from 24 h to 48 h after bleaching. In the 30-day recall, patients were also asked if they experienced pain during this 30-day period. As two bleaching sessions were performed, the VAS score obtained in both bleaching sessions was considered for statistical purposes. These values were computed for the maxillary arch.

ELIGIBILITY:
Inclusion Criteria:

The selected volunteers should:

* Present Good general state of health
* Be at least 18 years of age
* Have an acceptable oral hygiene
* Present the upper and lower arches without absence of teeth of first premolar right to the left first premolar.
* Have anterior teeth with any kind of restoration.
* Be No smoker
* Have the upper right canine with color 2M2 or darker

Exclusion Criteria:

The selected volunteers should not:

* Have medical history of diseases that can affect the results of the study
* Have made use of cigarettes in the last 30 days
* Have some important pathology in the oral cavity
* Be pregnant
* Be breastfeeding
* Have moderate advanced periodontal disease;
* Have consumed drugs, alcohol or any medication that can cover the results, as other types of anti-inflammatories or painkillers;
* Have used products indicated for dental sensitivity, as desensitizing toothpaste or similar product
* Present gingival recession
* Present exacerbated hypersensitivity history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tooth sensitivity | 1 hour after dental bleaching session
  Visual Analogic Scale (0-100) for Tooth Sensitivity.
Tooth sensitivity | 24 hours after dental bleaching session
  Visual Analogic Scale (0-100) for Tooth Sensitivity.
Tooth sensitivity | 48 hours after dental bleaching session
  Visual Analogic Scale (0-100) for Tooth Sensitivity.

SECONDARY OUTCOMES:
Subjective Color change | 30 days after dental bleaching session
  Subjective color evaluation comparing tooth color against a comercial color scale from A1 to D4
Objective Color change | 30 days after dental bleaching session
  Objective color evaluation using a spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: Marcos O Barceleiro, PhD, Principal Investigator — Full Professor
Locations (1):
- Universidade Federal Fluminense - School of Dentistry, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey CM. Tooth whitening: what we now know. J Evid Based Dent Pract. 2014 Jun;14 Suppl:70-6. doi: 10.1016/j.jebdp.2014.02.006. Epub 2014 Feb 13. PMID 24929591
- [Background] de Paula EA, Loguercio AD, Fernandes D, Kossatz S, Reis A. Perioperative use of an anti-inflammatory drug on tooth sensitivity caused by in-office bleaching: a randomized, triple-blind clinical trial. Clin Oral Investig. 2013 Dec;17(9):2091-7. doi: 10.1007/s00784-013-0918-2. Epub 2013 Jan 31. PMID 23371755
- [Background] de Paula EA, Nava JA, Rosso C, Benazzi CM, Fernandes KT, Kossatz S, Loguercio AD, Reis A. In-office bleaching with a two- and seven-day intervals between clinical sessions: A randomized clinical trial on tooth sensitivity. J Dent. 2015 Apr;43(4):424-9. doi: 10.1016/j.jdent.2014.09.009. Epub 2014 Sep 23. PMID 25257824
- [Background] Rezende M, Bonafe E, Vochikovski L, Farago PV, Loguercio AD, Reis A, Kossatz S. Pre- and postoperative dexamethasone does not reduce bleaching-induced tooth sensitivity: A randomized, triple-masked clinical trial. J Am Dent Assoc. 2016 Jan;147(1):41-9. doi: 10.1016/j.adaj.2015.07.003. Epub 2015 Nov 6. PMID 26562735
- [Background] da Costa Poubel LA, de Gouvea CVD, Calazans FS, Dip EC, Alves WV, Marins SS, Barcelos R, Barceleiro MO. Pre-operative use of dexamethasone does not reduce incidence or intensity of bleaching-induced tooth sensitivity. A triple-blind, parallel-design, randomized clinical trial. Clin Oral Investig. 2019 Jan;23(1):435-444. doi: 10.1007/s00784-018-2452-8. Epub 2018 Apr 25. PMID 29696420